CLINICAL TRIAL: NCT02778295
Title: Biomarker for Fabry Disease: BioFabry AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Patients With Fabry Disease (BioFabry)
Acronym: BioFabry
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BFA 06-2018
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Angiokeratomas; Chronic Kidney Disease; Ocular Abnormalities; Hearing Loss
Keywords: Fabry Disease; Biomarker
MeSH Terms: conditions — Angiokeratoma; Renal Insufficiency, Chronic; Hearing Loss; Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry, a blood sample will be taken via using a dry blood spot filter card. To proof the correct Fab-ry diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Fabry disease will be done.The analyses will done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Fabry disease or high-grade suspicion for Fabry disease

SUMMARY:
Development of a new mass spectrography-based biomarker for the early and sensitive diagnosis of Fabry disease from the blood

DETAILED DESCRIPTION:
Fabry disease is a progressive, inherited, multisystemic lysosomal storage disease characterized by specific neurological, cutaneous, renal, cardiovascular, cochleo-vestibular and cerebrovascular manifestations.

Annual incidence is reported to be 1 in 80,000 live births but this figure may underestimate disease prevalence. When late-onset variants of the disease are considered, a prevalence of approximately 1 in 3,000 has been suggested. Fabry disease is pan-ethnic.

Fabry disease is a disorder of glycosphingolipid metabolism caused by deficient or absent lysosomal alpha-galactosidase A activity related to mutations in the GLA gene (Xq21.3-q22) encoding the alpha-galactosidase A enzyme. Deficient activity results in accumulation of globotriaosylceramide (Gb3) within lysosomes, believed to trigger a cascade of cellular events.

Fabry disease is transmitted as an X-linked trait. The existence of atypical, late-onset, variants and the availability of specific therapy complicate genetic counseling.

The clinical picture covers a wide spectrum ranging from mild cases in heterozygous females, to severe cases in classically affected hemizygous males with no residual alpha-galactosidase A activity. These patients may have all the characteristic neurological (pain), cutaneous (angiokeratoma), renal (proteinuria, kidney failure), cardiovascular (cardiomyopathy, arrhythmia), cochleo-vestibular (hearing loss and vertigo) and cerebrovascular (transient ischemic attacks, strokes) symptoms of the disease.

Female patients may have very mild to severe symptoms. Pain is a common early symptom of Fabry disease (chronic pain characterized by burning and tingling paresthesia and occasional episodic crises characterized by agonizing burning pain). Pain may resolve in adulthood.

Anhidrosis or hypohidrosis may occur causing heat and exercise intolerance. Other signs include corneal changes ("cornea verticilata"), Definitive laboratory diagnosis involves demonstration of marked enzyme deficiency in hemizygous males. Enzyme analysis may occasionally help to detect heterozygotes but is often inconclusive due to random X-chromosomal inactivation, making molecular testing (genotyping) of females mandatory.

With age, progressive damage to vital organ systems develops, possibly leading to organ failure. End-stage renal disease and life-threatening cardiovascular or cerebrovascular complications limit the life-expectancy .

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 2 months
* The patient has a diagnosis of Fabry disease or a high-grade suspicion for Fabry disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

  * Positive family anamnesis for Fabry disease
  * Pin and burning in the hands and feet
  * Angiokeratomas
  * Gastrointestinal problems
  * Heart problems
  * Kidney problems

EXCLUSION CRITERIA:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of Fabry disease or no valid criteria for profound suspicion of Fabry disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Fabry disease or high-grade suspicion for Fabry disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Fabry disease related gene | 4 weeks
  Next-Generation Sequencing (NGS) of the GLA gene will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Fabry disease specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (3):
- Centogene GmbH, Rostock, Germany
- NIRMAN-University of Mumbai-Institute of Research in Mental and Neurological handicap, Mumbai, India
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided